CLINICAL TRIAL: NCT01790672
Title: Hydroxytyrosol as an Endogenous and Natural Antioxidant: Modulation by Alcohol Intake. Substudy 2. To Establish the Contribution of Wine Components on Hydroxytyrosol Body Concentrations and Biological Effects
Brief Title: Contribution of Wine Components on Hydroxytyrosol Body Concentrations and Biological Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Fundacion IMIM (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Hydroxytyrosol/FIS/2
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Contribution of Wine Components in Hydroxytyrosol Formation
Keywords: Antioxidants; Central Nervous System Agents; Wine
MeSH Terms: interventions — Ethanol; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Water (Placebo Comparator): Lemon-flavored water. 293 ml in pilot A, 147 ml in pilot B, 235 ml in pilot C, 147 ml in the definitive study.
  Interventions: Other: Water
- Alcoholized wine (Active Comparator): Wine 13º in pilot A (293 ml), B (147 ml) and the definitive study (147 ml). Corresponding to 30 g of ethanol in pilot A, 15 g of ethanol in pilot B and 15 g of ethanol in the definitive study.
  Wine 8º in pilot C (235 ml). Corresponding to 15 g of ethanol.
  Interventions: Dietary Supplement: Alcoholized wine
- De-alcoholized wine (Placebo Comparator): Wine 0º. Pilot A: 293ml; pilot B: 147 ml; pilot C: 235 ml; definitive study: 147 ml. Corresponding to 0 g of ethanol.
  Interventions: Dietary Supplement: De-alcoholized wine
- Ethanol (Active Comparator): Ethanol 13º in pilot A (293 ml), B (147 ml) and definitive study (147 ml). Corresponding to 30 g of ethanol in pilot A, 15 g of ethanol in pilot B and in the definitive study.
  Ethanol 8º in pilot C (235 ml). Corresponding to 15 g of ethanol.
  Ethanol was administered as a single dose of Vodka Absolut (40º) diluted in lemon-flavored water.
  Interventions: Dietary Supplement: Ethanol

INTERVENTIONS:
Dietary Supplement: Ethanol — Vodka Absolut
  Arms: Ethanol
Other: Water — Lemon-flavored water
  Arms: Water
Dietary Supplement: Alcoholized wine — Wine 13º or wine 8º
  Arms: Alcoholized wine
Dietary Supplement: De-alcoholized wine — Wine 0º
  Arms: De-alcoholized wine

SUMMARY:
The study is aimed at establishing the contribution of wine components on hydroxytyrosol body concentrations and biological effects.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting the study procedures and signing the informed consent.
* Male and female volunteers aged 18 to 55 years. No fixed sex ratio has been established.
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* The body mass index (BMI=weigh/height2) will range from 19 to 25 kg/m2, and the weight from 50 to 100 kg. 25-27 could be accepted.
* Women with regular menstrual cycle of 26-32 days.
* Subjects socially drinking and who had ingested wine at least once.

Exclusion Criteria:

* Not meeting the inclusion criteria.
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* History or clinical evidence of psychiatric disorders, alcoholism, drug abuse, or regular use of psychoactive drugs.
* Blood donation in the previous 8 weeks or participation in other clinical trials with drugs in the previous 12 weeks.
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* Subjects with intolerance or serious adverse reactions to ethanol.
* Regular use of any drug in the month prior to the study sessions, except for vitamins or diet supplements, that, in the opinion of the principal investigator or co-investigators designated by him, do not involve a risk for the subject and do not interfere with the study objectives. In this case they should be discontinued from one week before the experimental sessions to the end of them. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Taking more than 20 g of alcohol a day in women and more than 30 g in men.
* Taking more than 5 coffees, teas, cola drinks or other stimulating drinks or with xanthines daily in the 3 months prior to the study start.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Smokers or ex-smokers of less than one year.
* Subjects with positive serology to Hepatitis B, C or HIV.
* Pregnant or nursing women or positive pregnancy test in urine. Women not undertaking to follow reliable contraceptive measures during the study (such as abstinence, hormonal contraceptives, intrauterine devices, double-barrier methods or vasectomised partner).
* Women with amenorrhea or premenstrual syndrome of moderate or severe intensity.
* Nonsteroidal anti-inflammatory drugs, antioxidants or vitamins consumption in the last 2 weeks.
* Total cholesterol >6.00 mmol/l (240 mg/dl) or triglycerides >2.26 mmol/l (200 mg/dl).
* Vegetarians or subjects following aberrant diets.
* Physical exercise of >2h/day or >3000 kcal /week.

To be eligible, the subjects must agree to follow a poor polyphenols diet in the 72 hours prior to the start of each session and until 24 hours after.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Hydroxytyrosol biological fluids concentrations | 0-24h after administration
  Hydroxytyrosol concentrations in plasma and urine

SECONDARY OUTCOMES:
Ethanol concentration | 0-6h after administration
  Ethanol blood concentrations
Subjective drunkenness | 0-6h after administration
  Ethanol subjective effects measured using a visual analog scale
Vital signs | 0-24h after administration
  Blood pressure, oral temperature and heart rate
Ethanol metabolites concentrations | 0-24h after administration
  Ethanol metabolites recovery in urine
Dopamine metabolites concentrations | 0-24h after administration
  Dopamine metabolites recovery in urine
Oxidation biomarkers of proteins and lipids | 0-24h after administration
Psychomotor performance (DSST) | 0-6h after administration
  Psychomotor performance assessed by means of Digit symbol substitution test (DSST)
Gene expression of genes related with receptors and regulators/oxidative stress and antioxidant defence | Baseline
Platelets monoamine oxidase-B activity | Baseline
Breath ethanol | 30 min after administration
  Breath ethanol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Magí Farré, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut Mar, Barcelona, Barcelona, Spain